CLINICAL TRIAL: NCT03542578
Title: Diagnosis of Fatty Liver with Outpatient Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Achuthan Sourianarayanane, Asst Professor, Medical College of Wisconsin
Other Study IDs: PRO00029401
Record Dates: First submitted 2018-04-24; First posted 2018-05-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Liver Steatoses
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: outpatient evaluation of fatty liver — outcome of ultrasound evaluation of liver in clinical outpatient settings

SUMMARY:
This study will evaluate whether ultrasound performed during outpatient visit is effective in early diagnosis of fatty liver.

DETAILED DESCRIPTION:
All patients presenting to dedicated hepatology clinic with concern for fatty liver will be evaluated by ultrasound. This will be compared with standard imaging performed for this condition. The data will be compared for effectiveness of outpatient evaluation with dedicated imaging currently practiced

ELIGIBILITY:
Inclusion Criteria:

* all patients presenting to dedicated clinic

Exclusion Criteria:

* presence of ascites, inability to give consent to have study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting outpatient clinic will be evaluated
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Outpatient ultrasound in diagnosis of fatty liver diagnosis | Bedside evaluation performed after consent and compared with radiological imaging perfomed within 3 months of this bedside evaluation
  Effectiveness of outpatient evaluation by outpatient bedside ultrasound device in diagnosis of fatty liver compared to standard radiological evaluation. Comparing presence and severity of steatosis reported by standard radiological imaging with bed side imaging tool.

CONTACTS AND LOCATIONS:
Overall Officials: Achuthan Sourianarayanane, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No